CLINICAL TRIAL: NCT02709174
Title: Diagnosing Pulmonary Embolism in Pregnancy: Are Biomarkers and Clinical Prediction Models Useful?
Brief Title: Pulmonary Embolism in Pregnancy: Biomarkers and Clinical Predictive Models
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 5699
Record Dates: First submitted 2015-08-19; First posted 2016-03-15 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2016-03

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Pregnancy; D-Dimer
MeSH Terms: conditions — Pulmonary Embolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pregnant with pulmonary embolism: Pregnant women who underwent diagnostic imaging to evaluate for suspected PE at our institution
  Interventions: Procedure: blood draw
- pregnant without pulmonary embolism: Pregnant women who underwent diagnostic imaging to evaluate for suspected PE at our institution

INTERVENTIONS:
Procedure: blood draw — blood draw
  Groups: pregnant with pulmonary embolism

SUMMARY:
Objective: To evaluate whether trimester specific d-dimer levels and brain natriuretic protein (BNP), along with the modified Wells score (MWS), is a useful risk stratification tool to exclude pregnant women at low-risk of pulmonary embolism (PE) from diagnostic imaging with radiation exposure.

DETAILED DESCRIPTION:
To account for all women meeting the study eligibility criteria, this study utilized a combined prospective and retrospective arm. Pregnant women who underwent diagnostic imaging to evaluate for suspected PE at our institution were prospectively enrolled from February 2014 to August 2015. Both d-dimer and BNP serum levels were drawn, and a MWS was assigned. All pregnant women diagnosed with a PE that underwent diagnostic imaging and had a d-dimer level drawn from January 2009 to June 2014 were retrospectively enrolled. Patient electronic records were used to apply the MWS and analyze their risk.

ELIGIBILITY:
Inclusion criteria:

* adult pregnant women >= 18 years old
* d-dimer obtained and if the patient was pregnant at the time of PE diagnosis
* patient presented to the Emergency Department or Labor and Delivery unit
* patient presented with signs and symptoms suspicious for PE

Exclusion criteria:

* non-pregnant patients
* patients < 18 years old

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women who presented to the Emergency Department or Labor and Delivery unit with signs and symptoms suspicious for PE
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Serum D-dimer levels (ug/ml) | 18 months
  Trimester specific D-dimer levels to identify pregnant women at low risk for pulmonary embolism, thereby avoiding radiation exposure

SECONDARY OUTCOMES:
Modified Well's Criteria- a risk scoring system for likelihood of pulmonary embolism | 18 months
  A Modified Wells score of >4 suggests pulmonary embolism is likely and therefore diagnostic imaging needed

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Parilla, MD, Principal Investigator — Advocate Health